CLINICAL TRIAL: NCT05856331
Title: Phase 2, Double-Blind, Randomized, Active-Control, Parallel Group Study to Assess the Pharmacokinetics, Pharmacodynamics, Immunogenicity, and Safety of SAR447537 (INBRX-101) Compared to Plasma-Derived Alpha1-Proteinase Inhibitor (A1PI) Augmentation Therapy in Adults With Alpha-1 Antitrypsin Deficiency (AATD) Emphysema
Brief Title: Study of SAR447537 (INBRX-101) Compared to Plasma-derived A1PI Therapy in Adults With AATD Emphysema
Acronym: ELEVAATE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INBRX101-01-201; 2023-508084-76-00 (Registry Identifier: CTIS)
Record Dates: First submitted 2023-03-28; First posted 2023-05-12 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Alpha 1-Antitrypsin Deficiency; Emphysema
Keywords: AATD; Alpha 1-Antitrypsin Deficiency; Emphysema; SAR447537; INBRX-101; A1PI; AAT
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency; Emphysema | interventions — alpha 1-Antitrypsin; Respreeza

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized, active-control, parallel group interventional study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SAR447537 (INBRX-101) Q3W (Experimental): IV every 3-weeks (Q3W) and placebo (normal saline)
  Interventions: Drug: SAR447537
- SAR447537 (INBRX-101) Q4W (Experimental): IV every 4-weeks (Q4W) and placebo (normal saline)
  Interventions: Drug: SAR447537
- Zemaira (A1PI) (Active Comparator): 60 mg/kg IV once weekly (QW) and placebo (normal saline)
  Interventions: Drug: Zemaira

INTERVENTIONS:
Drug: SAR447537 — A1PI, Recombinant, Bivalent Fc Fusion Protein
  Arms: SAR447537 (INBRX-101) Q3W; SAR447537 (INBRX-101) Q4W
Drug: Zemaira — Alpha1-Proteinase Inhibitor (Human)
  Other Names: Respreeza
  Arms: Zemaira (A1PI)

SUMMARY:
Phase 2 study to compare SAR447537 (INBRX-101) to plasma derived A1PI therapy in adults with AATD emphysema

DETAILED DESCRIPTION:
This is a Phase 2, Double-Blind, Randomized, Active-Control, Parallel Group Study to Assess the Pharmacokinetics, Pharmacodynamics, Immunogenicity, and Safety of SAR447537 (INBRX-101) Compared to Plasma-Derived Alpha1-Proteinase Inhibitor (A1PI) Augmentation Therapy in Adults With Alpha-1 Antitrypsin Deficiency (AATD) Emphysema.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females 18-80 years of age, inclusive, at the time of screening
2. Diagnosis of AATD
3. Evidence of emphysema secondary to AATD
4. FEV1 of ≥ 30% and ≤ 80% predicted at screening
5. Current non-smoking status.

Exclusion Criteria:

1. Receipt of A1PI augmentation therapy within 5 weeks prior to the first dose of study drug
2. Known or suspected allergy to components of SAR447537 (INBRX-101), A1PI or human IgG
3. Known selective or severe Immunoglobulin A (IgA) deficiency
4. Known or suspected diagnosis of type 1 diabetes or diagnosed with uncontrolled type 2 diabetes
5. Received IV immunoglobulins, monoclonal antibodies and/or other biologic therapies within 30 days
6. On waiting list for lung or liver transplant
7. Acute respiratory tract infection or COPD exacerbation within 4 weeks prior to or during screening
8. Evidence of decompensated cirrhosis
9. Active cancers or has a history of malignancy within 5 years prior to screening
10. History of unstable cor pulmonale
11. Clinically significant congestive heart failure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2023-10-12 (Actual); Primary Completion 2025-08-06 (Actual); Study Completion 2025-08-06 (Actual)

PRIMARY OUTCOMES:
Serum functional AAT (fAAT) levels at steady-state | 32 Weeks
  To assess the mean change in average fAAT concentration as measured by anti-neutrophil elastase capacity [ANEC] from baseline to average serum trough fAAT concentration at steady-state (Ctrough,ss) in participants treated with SAR447537 compared to A1PI

SECONDARY OUTCOMES:
fAAT Concentration changes | 32 Weeks
  Mean change in serum fAAT concentration from baseline to fAAT average concentration at steady-state (Cavg, ss) in participants treated with SAR447537 compared to A1PI.
Days with fAAT above the lower limit of the normal range | 32 weeks
  Percentage of days with fAAT above the lower limit of the normal range during steady-state dosing in participants treated with SAR447537 compared to A1PI.
Incidence of TEAEs | 32 Weeks
  Incidence of all treatment-emergent adverse events (TEAEs), TEAEs ≥ Grade 3, serious adverse events (SAEs), TEAEs leading to IMP discontinuation, adverse events of special interest (AESI) (including infusion- related reactions).
Anti-drug antibodies | 32 Weeks
  Frequency of anti-drug antibodies (ADA) against SAR447537 and endogenous AAT, as well as neutralizing ADA (NAb) against SAR447537 and endogenous AAT.
Population Pharmacokinetics: Clearance | 32 Weeks
  Modeling by means of appropriate software to characterize the pharmacokinetic profile of SAR447537 via estimation of the parameter clearance
Population Pharmacokinetics: Volume of Distribution | 32 Weeks
  Modeling by means of appropriate software to characterize the pharmacokinetic profile of SAR447537 via estimation of the parameter volume of distribution
Covariate Analysis: Biometric Values: Weight | 32 Weeks
  Assessment of the impact of participant's weight [in kg] on the pharmacokinetic profile of SAR447537
Covariate Analysis: Biometric Values: Height | 32 Weeks
  Assessment of the impact of participant's height [in cm] on the pharmacokinetic profile of SAR447537
Covariate Analysis: Biometric Values: Age | 32 Weeks
  Assessment of the impact of participant's age [in years] on the pharmacokinetic profile of SAR447537
Covariate Analysis: Biometric Values: Sex | 32 Weeks
  Assessment of the impact of participant's sex [male or female] on the pharmacokinetic profile of SAR447537

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (65):
- United States (39):
  - University of Alabama at Birmingham- Site Number : 105, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - St Joseph's Hospital and Medical Center- Site Number : 126, Phoenix, Arizona
  - St Joseph's Hospital and Medical Center, Phoenix, Arizona
  - David Geffen School of Medicine- Site Number : 124, Los Angeles, California
  - David Geffen School of Medicine, Los Angeles, California
  - UC Davis Comprehensive Cancer Center- Site Number : 110, Sacramento, California
  - UC Davis Medical Center, Sacramento, California
  - National Jewish Medical and Research Center- Site Number : 123, Denver, Colorado
  - National Jewish Medical and Research Center, Denver, Colorado
  - Western Connecticut Medical Group, Danbury, Connecticut
  - University of Florida College of Medicine- Site Number : 101, Gainesville, Florida
  - University of Florida, Gainesville, Florida
  - Bruce W. Carter Miami VA Medical Center - NAVREF - PPDS- Site Number : 114, Miami, Florida
  - University of Miami, Miami, Florida
  - Pulmonary and Sleep of Tampa Bay- Site Number : 115, Tampa, Florida
  - Pulmonary and Sleep of Tampa Bay, Tampa, Florida
  - Loyola University Medical Center- Site Number : 112, Maywood, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Indiana University, Indianapolis, Indiana
  - M Health Fairview Clinics and Surgery Center - Minneapolis- Site Number : 125, Minneapolis, Minnesota
  - M Health Fairview Clinics and Surgery Center - Minneapolis, Minneapolis, Minnesota
  - Hannibal Regional Healthcare System-HRMG-Hannibal- Site Number : 111, Hannibal, Missouri
  - Hannibal Clinic, Hannibal, Missouri
  - Columbia University Irving Medical Center- Site Number : 104, New York, New York
  - Oregon Health and Science University- Site Number : 117, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Clinical Research Associates Of Central PA , LLC- Site Number : 128, DuBois, Pennsylvania
  - Clinical Research Associates Of Central PA , LLC, DuBois, Pennsylvania
  - Penn State Health Milton S. Hershey Medical Center- Site Number : 122, Hershey, Pennsylvania
  - Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Temple University Hospital- Site Number : 130, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Velocity Clinical Research - Spartanburg - PPDS- Site Number : 120, Spartanburg, South Carolina
  - Velocity Clinical Research - Spartanburg - PPDS, Spartanburg, South Carolina
  - Houston Methodist Hospital- Site Number : 113, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - University of Utah Health, Salt Lake City, Utah
  - University of Utah Health Care- Site Number : 106, Salt Lake City, Utah
- Australia (11):
  - Donna McIntyre, Brisbane, Queensland
  - Queensland Centre for Pulmonary Transplantation, Chermside, Queensland
  - Royal Adelaide Hospital, North Adelaide, South Australia
  - Eastern Health Clinical School, Box Hill, Victoria
  - Investigational Site Number : 203, Fitzroy, Victoria
  - St Vincent Hospital Melbourne, Fitzroy, Victoria
  - Frankston Hospital, Frankston, Victoria
  - Institute for Respiratory Health, Nedlands, Western Australia
  - Investigational Site Number : 206, Nedlands, Western Australia
  - Investigational Site Number : 201, Adelaide
  - Investigational Site Number : 202, Chermside
- Denmark (2):
  - Investigational Site Number : 701, Hellerup
  - Investigational Site Number : 702, Vejle
- New Zealand (4):
  - NZRSI, Greenlane, Auckland
  - Investigational Site Number : 403, Auckland
  - Investigational Site Number : 404, Wellington
  - P3 Research, Wellington
- Poland (2):
  - Investigational Site Number : 801, Warsaw, Masovian Voivodeship
  - Investigational Site Number : 802, Krakow
- Spain (2):
  - Investigational Site Number : 901, Santander, Cantabria
  - Investigational Site Number : 903, Santiago de Compostela, La Coruña
- Investigational Site Number : 601, Gothenburg, Sweden
- United Kingdom (4):
  - Ninewells Hospital - PPDS, Dundee, Angus
  - Investigational Site Number : 306, Wythenshawe, Cheshire West And Chester
  - Medicines Evaluation Unit, Manchester, Cheshire
  - Investigational Site Number : 302, Birmingham, Warwickshire

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org